CLINICAL TRIAL: NCT06618014
Title: A Single-Arm Phase II Trial of Neoadjuvant Toripalimab, Docetaxel, Plus Carboplatin in Patients With Localized Triple-Negative Breast Cancer
Brief Title: Neoadjuvant Toripalimab Plus Docetaxel and Carboplatin in Patients With Localized TNBC (NeoTOP)
Acronym: NeoTOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoTOP
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: TNBC, neoadjuvant, immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — toripalimab; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant TCb+Toripalimab (Experimental): Patients receive toripalimab (240 mg) plus docetaxel and carboplatin (AUC=4) on day 1 of each 21-day cycle for 6 cycles.
  Interventions: Drug: Toripalimab; Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Toripalimab — Toripalimab was given 240 mg intravenously on day 1 of each 21-day cycle for 6 cycles.
Drug: Docetaxel — Docetaxel was administered at a dose of 75 mg/m2 on day 1 of each 21-day cycle for 6 cycles.
Drug: Carboplatin — Carboplatin was given dosed to an area under the serum concentration-time curve (AUC) of 4 on day 1 of each 21-day cycle for 6 cycles.

SUMMARY:
This study aims to investigate efficacy and safety of neoadjuvant toripalimab plus docetaxel and carboplatin in patients with localized triple-negative breast cancer.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy combined with immunotherapy is the recommended therapeutic approach for patients with localized triple-negative breast cancer (TNBC). The combination regimen improved the pCR rate of triple negative breast cancer, but its side effects also increased. In the KEYNOTE-522 trial, 78% of patients receiving pembrolizumab combined with anthracycline and paclitaxel chemotherapy experienced grade 3 or higher adverse reactions, while the incidence of grade 3 or higher adverse events for patients receiving tislelizumab plus nab-paclitaxel and carboplatin in the CTRIO study was 53.2%. Toripalimab (an anti PD-1 monoclonal) combined with paclitaxel (albumin binding type) for first-line treatment of recurrent or metastatic TNBC was recently approved based on the results from the TORCHLIGHT study. This study aims to investigate efficacy and safety of neoadjuvant toripalimab plus docetaxel and carboplatin in patients with localized TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed TNBC. ER and PR negatives are defined as < 10% of cells expressing hormone receptors by IHC analysis. HER2 negative is defined as IHC 0 or 1+, or ISH-negative.
* Treatment-naive clinical stage T1-4N1-N3 or T2-4N0 localized TNBC.
* Female patients aged ≥18 years, < 70 years.
* Able to comply with the required protocol and follow-up procedures.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy ≥12 weeks.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥90 x 109/L, and Hemoglobin ≥90 g/L (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 1.5 x ULN.
* Adequate renal function: Serum creatinine ≤ 1.5 x ULN, and creatinine clearance ≥ 50 ml/min.
* Subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Inflammatory breast cancer or stage IV breast cancer.
* Prior systemic antitumor treatment for any malignancy, including chemotherapy, radiotherapy, immunotherapy and targeted therapy.
* History of another malignancy in the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Inability to comply with protocol or study procedures.
* Subjects with active, known or suspected autoimmune disease. Subjects in conditions not expected to recur in the absence of an external trigger, or not requiring systemic treatment are permitted to enroll.
* Previous history of interstitial lung disease/pneumonia.
* Patient who has had an allogeneic tissue/solid organ transplant.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Patient who has active serious infection (e.g. pyrexia of or 38.0℃ over)
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Women who are pregnant or nursing.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | 1 week after surgery
  The number of patients with pCR out of the total number of participants using a definition of ypT0/Tis ypN0 after neoadjuvant therapy and surgery.

SECONDARY OUTCOMES:
Rate of Residual Cancer Burden (RCB) of 0-1 | 1 year
  The number of patients with RCB of 0-1 after neoadjuvant therapy and surgery.
Objective Response Rate (ORR) | 1 year
  The number of patients with complete response and partial response out of the total number of participants.
Event-Free Survival (EFS) | 3 years after the last patient is enrolled
  EFS was defined as the time from registration to disease progression (local relapse or distant metastases) or death from any cause, whichever came first.
Safety of the combination therapy | 1 year
  Adverse events (AEs) were graded according to NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Tang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan (SAP) will be shared with other researchers after publication of the study.
Supporting Information: Study Protocol, SAP
Time Frame: Study Protocol and Statistical Analysis Plan (SAP) will be shared with other researchers after publication of the study.